CLINICAL TRIAL: NCT00501566
Title: SR121463B in Cirrhotic Ascites Treatment With Normonatraemia: A Placebo-Controlled, Dose-Comparison Study
Brief Title: Satavaptan Dose-Ranging Study in Normonatraemic Patients With Cirrhotic Ascites
Acronym: Normo~CAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI5563; SR121463
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Ascites; Liver Cirrhosis
Keywords: cirrhotic ascites
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — satavaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: satavaptan (SR121463B)

SUMMARY:
The primary objective is to determine the optimal dose or range of doses of SR121463B for the treatment of ascites when used concomitantly with a standard dose regimen of spironolactone and furosemide.

The secondary objective is to determine the tolerability of different fixed doses of SR121463B over a 14 day treatment period in cirrhotic ascites.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of the liver confirmed by ultrasound, endoscopic examination or biochemical evidence
* Moderate or tense ascites
* Serum sodium of >130 mmol/l.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2004-04; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight | within 14 days

SECONDARY OUTCOMES:
Abdominal girth and discomfort | 14 days
Paracentesis | 14 days
Quality of life | 14 days

CONTACTS AND LOCATIONS:
Locations (12):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com